CLINICAL TRIAL: NCT03989856
Title: Effect of Laparoscopic Suturing Versus Bipolar Coagulation on Ovarian Reserve in Patients Undergoing Endometriotic Ovarian Cystectomy.
Acronym: Eolsb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed abd elfatah elsenity, Lecturer of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 123456789
Record Dates: First submitted 2019-06-15; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Ovary Injury
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: The study population comprises females in childbearing period underwent laparoscopic ovarian cystectomy at Ain Shams University Maternity Hospital, Obstetric and Gynecology Department, Faculty of medicine.
Who Masked: Participant, Investigator
Masking Description: Allocation and concealment will be done by sequentially sealed opaque envelopes. 60 envelopes will be numbered serially from 1 to 60, 30 envelopes will contain the letter c and the other 30 will contain the letter S.
  In each envelope, the corresponding letter which donates the allocated group will be put according to the randomization table and them all envelopes will be closed and put in one box. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suturing group (Experimental): The sutures will be performed with intracorporeal knots using 2-0 polyglican absorbable sutures (Vicryl; Ethicon Inc., New Jersey, USA). Suture is performed using needle holders for the closure of ovarian parenchyma and controlling bleeding. Bleeding from ovarian hilus will only resolve by suturing.
  The running suture starting from central area, around the ovarian hilus to peripheral tissue, will be performed with intraovarian knots to re-approximate the edges to achieve satisfying hemostasis. Knots will not be detectable on the ovarian surface for prevention of adhesion. Mean time for hemostasis of ovary was recorded in a form. The cyst wall will be removed from the abdomen by means of an endobag. All resected cyst walls will be sent to the pathology laboratory, to confirm the histopathology of endometriosis.
  Interventions: Device: 2-0 polyglican absorbable sutures
- Bipolar group (Active Comparator): In bipolar coagulation group, after stripping the ovarian cyst wall, bipolar coagulation technique will be used to control significant bleeding (40 W current; Richard Wolf, Germany). In laparoscopic suturing group, no bipolar coagulation will be performed during or after stripping the ovarian cyst wall.
  Interventions: Device: Diathermy

INTERVENTIONS:
Device: 2-0 polyglican absorbable sutures — The sutures will be performed with intracorporeal knots using 2-0 polyglican absorbable sutures (Vicryl; Ethicon Inc., New Jersey, USA). Suture is performed using needle holders for the closure of ovarian parenchyma and controlling bleeding. Bleeding from ovarian hilus will only resolve by suturing.
  Arms: Suturing group
Device: Diathermy — bipolar coagulation technique will be used to control significant bleeding (40 W current; Richard Wolf, Germany). I
  Arms: Bipolar group

SUMMARY:
In women undergoing laparoscopic ovarian cystectomy which is less harmfull on the ovarian reserve (electrocoagulation or suturing).

DETAILED DESCRIPTION:
The aim of the present study was to determine which hemostatic procedure (hemostatic suture or electrocautery) may be less harmful after laparoscopic cystectomy, based on the longterm status of the ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 45.
2. Regular menstrual cycle.
3. Unilateral ovarian cyst clinical & us finding as endometriotic cyst.
4. C/O of pelvic pain.
5. No medications (oral pills & hormonal drugs) in the past 3 monthes before enrollement.
6. No evidence of endocrine disorders (DM, Thyroid dysfunction,hyper prolactenemia, congenital adrenal hyperplesia, cushing's syndrome or adrenal insufficiency)
7. No previous adnexial surgery.
8. Pathology diagnosis of excised ovarian tissue (endometriotic cyst)
9. Appropriate medical condition for laparoscopic surgery.
10. Completely understand the process of the study with written consent.

Exclusion Criteria:

1. PCO according to Rotterdam criteria.
2. Pathological diagnosis of excised ovarian tissue as non endometriotic cyst.
3. Previous ovarian surgery.
4. Suspected ovarian malignancy.
5. Patient whose histopathology showed benign cyst apart from endometrioma.
6. Irregular menstrual cycles.
7. Post menopausal status.
8. Bilateral ovarian cyst.
9. AMH < 0.5 ng/ml.
10. Premature ovarian failure in family.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve | 3 months
  By measuring Anti-mullerian hormone

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd elfattah elsenitt, Lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams maternity teaching hospital, Cairo, Abbasia, Egypt